CLINICAL TRIAL: NCT06284538
Title: Randomized Controlled Study to Evaluate the Performance and Safety of a Linear Hyaluronic Acid-based Medical Device in the Treatment of Wounds
Brief Title: Study to Evaluate the Effectiveness of a Medical Device Based on Hyaluronic Acid in Wounds
Acronym: WOUND-H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Argentia S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA-01-23
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Wound Healing Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WOUND-H (Experimental): STUDY FOR THE ASSESSMENT OF THE EFFECTIVENESS OF A MEDICAL DEVICE BASED ON HYALURONIC ACID IN WOUNDS
  Interventions: Device: NOVA.EMOSTOP RE-EPITHELIZING
- Braccio controllo (Active Comparator): NORMAL STANDARD THERAPIES FOR WOUND TREATMENT (CLEANING AND DISINFECTION)
  Interventions: Device: NOVA.EMOSTOP RE-EPITHELIZING

INTERVENTIONS:
Device: NOVA.EMOSTOP RE-EPITHELIZING — RE-EPITHELIZING GEL BASED ON HYALURONIC ACID

SUMMARY:
The primary objective of the study is to evaluate the safety and performance of a Class IIB medical device based on linear hyaluronic acid used in the treatment of post-surgical wounds. The outcomes of the study are the improvement of wound healing assessed through the Clinical Healing score (score from 0 to 5), which includes the evaluation of: redness, edema, suppuration, healthy granulation tissue and signs of re-epithelialization; the percentage of patients with completely healed wounds at day 30 post-treatment; the pain perceived by the patient when changing the dressing; the frequency of adverse events.

DETAILED DESCRIPTION:
Wound healing is a complex and dynamic process, which is still far from being fully understood. Wounds can be classified based on different characteristics such as the triggering factor, exposure to the external environment, depth of the wound, healing time period, potential risk of infections1. Two main processes are involved in wound healing: regeneration and repair. Regeneration involves the activation of stem cells capable of reconstituting the integrity of the tissue which will be indistinguishable from the tissue before the injury. Many strategies and products have been proposed in order to improve wound healing, reduce pain and morbidity for patients such as wound dressing, growth factors, skin substitutes, collagen dressing, topical insulin , the antioxidant, the hyperbaric chamber, etc. Hyaluronic acid (HA) was discovered in 1934 by Meyer and Palmer in bovine ocular vitreous. It is a naturally occurring glycosaminoglycan that, by virtue of its viscosity, elasticity and other rheological properties, acts as an ocular lubricant and as a lubricating and shock-absorbing fluid in the joints. It is produced by fibroblasts within the cell membrane and then released into the extracellular space. Inside the skin, it plays an important role in hydrating the extracellular space; constitutes a matrix to support the normal functions of cells; it also has functions in space filling, lubrication, wound healing, modulation of inflammatory cells, and scavenging of free radicals. Due to its remarkable biomedical and tissue regeneration potential, HA is widely used in the treatment of wounds under different formulations such as gauzes, creams and gels4, showing significant clinical results.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with post-surgical wounds
* subjects capable of complying with the protocol procedures
* signing of informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* inadequate contraceptive procedures in fertile women
* chronic concomitant treatment with local antiseptics, use of anti-inflammatory drugs (steroids and non-steroids), analgesics, antineoplastics or immunosuppressants
* non-therapeutic use of psychoactive substances, drug and/or alcohol abuse
* immunodeficiencies (including HIV infection)
* Oncology patients;
* known allergies, hypersensitivity or intolerance to any of the substances administered in this study
* any medical or non-medical condition that may significantly reduce the possibility of obtaining reliable data and achieving the objectives of the study
* Participation in clinical trials with devices or drugs within 3 months prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
improvement in Clinical Healing score at visit 3 | 30 days
  improvement in Clinical Healing score at visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Loredana Comito, Monitor, Study Chair — Clinical Research Consulting S.r.l.
Locations (1):
- Casa di cura riabilitativa Villa Sofia, Acireale, Catania, Italy

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT06284538/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT06284538/ICF_001.pdf